CLINICAL TRIAL: NCT03861416
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled Study of the Safety and Efficacy of Unifuzol® in Patients With Peripheral Arterial Disease
Brief Title: "Unifuzol®" in Patients With Peripheral Arterial Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: POLYSAN Scientific & Technological Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNI-II-2016
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Arterial Occlusive Disease; intermittent claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Intermittent Claudication | interventions — Arginine; Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unifuzol® 1.4% 500 ml (Experimental): Patients receive the infusion of investigational drug L-arginine 1.4% 500 ml IV daily for 10 days
  Interventions: Drug: L-arginine 1.4% 500 ml
- Unifuzol® 1.4% 250 ml (Experimental): Patients receive the infusion of L-arginine 1.4% 250 ml + placebo 250 ml IV daily for 10 days
  Interventions: Drug: L-arginine 1.4% 250 ml + placebo 250 ml
- Placebo 500 ml (Placebo Comparator): Patients receive the infusion of placebo solution for intravenous infusions 500 ml IV daily for 10 days.
  Interventions: Drug: Placebo solution

INTERVENTIONS:
Drug: L-arginine 1.4% 500 ml — Infusion of L-arginine 1.4% solution by 500 ml (2 vials 250 ml each) IV daily for 10 days
  Other Names: Unifuzol® 1.4%
  Arms: Unifuzol® 1.4% 500 ml
Drug: L-arginine 1.4% 250 ml + placebo 250 ml — Infusion of L-arginine 1.4% solution 250 ml IV daily for 10 days and placebo infusion by 250 ml IV daily for 10 days.
  Other Names: Unifuzol® 1.4% 250 ml and placebo 250 ml
  Arms: Unifuzol® 1.4% 250 ml
Drug: Placebo solution — Infusion of Ringer's solution by 500 ml (2 vials 250 ml each) IV daily for 10 days
  Other Names: Ringer's solution
  Arms: Placebo 500 ml

SUMMARY:
The present study is a multicenter, randomized, double-blind, placebo-controlled study of the safety and efficacy of the drug Unifuzol® (L-arginine) in patients with obliterating atherosclerosis of the lower extremities. The study recruits patients 40-79 years old with a confirmed diagnosis of chronic ischemia of the lower limb and a stable symptom of intermittent claudication that occurs when walking a distance of 100-299 meters. L-arginine improves microcirculation due to activation of nitrogen monoxide production and stimulates capillary blood flow, thus can probably improve the quality of life of patients with intermittent claudication. The criterion for treatment efficacy will be an increase in the maximum walking distance measures before and on the next day after the end of treatment course.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Male and female patients 40-79 years old
3. Patients with atherosclerosis of native arteries of the lower extremity vessels (ICD-10 code: I70.2)
4. Clinical syndrome of chronic lower limb ischemia
5. The symptom of intermittent claudication persisting for 6 months or more (before the start of screening), causing a stable restriction of physical activity to the maximum walking distance 100-299 m
6. The ankle-brachial index (ABI) less than 0.9; in patients with diabetes mellitus ABI >1.2 is acceptable, provided the occlusion of the main arteries of the lower extremities is confirmed
7. Patient consent to the use of adequate methods of contraception or full abstinence from sexual activity for the period of the study and within 30 days after its completion
8. The difference between the maximum walking distance at the second and the first treadmill test at the screening (interval at least 3 days) does not exceed 25% from baseline, i.e. the first treadmill test
9. Patients not receiving drugs for the treatment of atherosclerosis obliterans of the lower extremities or receiving them in constant doses for at least 6 weeks prior to screening.
10. No contraindications for treadmill test

Exclusion Criteria:

1. Intolerance or hypersensitivity to the components of the study drug.
2. Intake of succinic acid, L-arginine, malic acid, fumaric acid, anticoagulants, or hormones (with the exception of insulin) within 6 weeks before the start of screening, or the use of these medications is scheduled within the patient's participation in the study
3. Any severe disease or condition that may make it unsafe and/or impossible for the patient to participate in the study and/or lead to the inability of the patient to comply with the study procedures (including, but not limited to: renal failure, hepatic failure, blood diseases, psychiatric conditions, infections)
4. History of malignancy (with the exception of basal cell skin cancer)
5. Alcohol or drug abuse
6. The presence of clinically significant decompensated cardiovascular diseases (unstable angina or stenocardia of functional class III and above, chronic heart failure III - IV class according to NYHA, uncontrolled arterial hypertension, acute cerebrovascular accident or acute myocardial infarction within 6 months prior to screening, unstable arrhythmias, deep venous thrombosis, stenosis of the internal carotid arteries >70%, aortic aneurysm)
7. Decompensation of the peripheral circulation: rest pain, trophic ulcers, gangrene
8. Any other diseases that affect the assessment of walking distance and limit patient's physical activity
9. The level of glycated hemoglobin (HbA1c) >= 8%
10. Planned reconstructive surgery on the limb vessels within 6 months from screening
11. Amputation on one or both limbs or planned amputation within 6 months from screening
12. Other circumstances impeding patient compliance with the schedule of procedures
13. For patients applying or planning the use of NSAIDs: the inability to cancel the use of NSAIDs 12 hours before the treadmill test.
14. The body mass index >35
15. Contraindications for conducting the treadmill test
16. Heart rate is more than 80% of the maximum frequency (the maximum frequency is defined as 220 - age) at the moment of pain in the legs.
17. Depression of an ST segment or the occurrence of sustained (lasting more than 30 seconds) cardiac rhythm or conduction disturbances during a treadmill test.
18. Drop of systolic blood pressure during the first 5 minutes after the completion of the treadmill test
19. Participation in another clinical study
20. Pregnancy or breastfeeding
21. Any other diseases / conditions in the stage of decompensation
22. Employees of the research center and their family members.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-10-26 (Actual)

PRIMARY OUTCOMES:
Maximum walking distance | day 11, day 30
  The change in the maximum walking distance on the next day (day 11) after the completion of treatment course and on day 30 in comparison with the initial value. The change will be expressed as the ratio of the natural logarithms of the maximum walking distance on day 11 and to the baseline value (day 1).

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail S Bogomolov, MD, PhD, Study Director — St. Petersburg State Medical University n.a. I.P.Pavlov
Locations (19):
- Russia (19):
  - Regional Clinical Hospital, Barnaul
  - Kursk City Clinical Emergency Hospital, Kursk
  - City Clinical Hospital № 15 named O.M. Filatov, Moscow
  - Medical and sanitary Department of the Ministry of Internal Affairs of the Russian Federation in Moscow, Moscow
  - City Clinical Hospital №2 of the Novosibirsk Region, Novosibirsk
  - National Medical Research Center named after Academician E.N. Meshalkin, Novosibirsk
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
  - Multidisciplinary center of modern medicine "Euromed", Omsk
  - Orenburg Regional Clinical Hospital, Orenburg
  - Rostov State Medical University, Rostov-on-Don
  - Ryazan Regional Clinical Cardiological dispensary, Ryazan
  - City General Hospital №2, Saint Petersburg
  - City Hospital №38 named after N.A. Semashko, Saint Petersburg
  - Consultative and diagnostic center No. 85, Saint Petersburg
  - Road Clinical Hospital of the Russian Railways Open Joint-Stock Company, Saint Petersburg
  - St. Petersburg State Medical University n.a. I.P.Pavlov, Saint Petersburg
  - Regional Clinical Cardiology Dispensary, Saratov
  - Clinical hospital №10 of the Yaroslavl region, Yaroslavl
  - Regional Clinical Hospital of the Yaroslavl region, Yaroslavl